CLINICAL TRIAL: NCT06822894
Title: Clinical Implications of Three-vessel Ultrasonic Flow Ratio Measurement in Patients With Coronary Artery Disease
Acronym: FUNCTION III
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-2-4034
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease (CAD)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not applicable- observational study — UFR is a novel IVUS-derived modality for fast computation of FFR without pressure wires and adenosine

SUMMARY:
This is a prospective, observational, single-center study. The main purpose of this study is to explore the predictive value of three coronary vessel-ultrasonic flow ratio (3V-UFR) for major adverse cardiovascular events (MACE) in patients with coronary artery disease within one year. The study will be conducted in Fuwai Hospital, and a total of at least 494 patients with all the three coronary vessel diameter stenoses ≥30% are planned to be recruited. Participants who meet the inclusion criteria and do not meet the exclusion criteria will undergo intravascular ultrasound (IVUS). IVUS imaging will be sent to an independent core laboratory for offline UFR calculation. Subsequently, a one-year follow-up was conducted on the patients. The primary endpoint was MACE within one year, which included cardiac death, any myocardial infarction, and ischemia-driven coronary revascularization. The association between the 3V-UFR (low 3V-UFR and high 3V-UFR grouped by median of 3V-UFR) and MACE is investigated, to determine its role in clinical prognosis for patient with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina pectoris, unstable angina pectoris, or after the acute phase of myocardial infarction
* Age ≥18 years
* Written informed consent
* Angiographically confirmed ≥30% diameter stenosis in all three major epicardial coronary arteries (left anterior descending, left circumflex, and right coronary artery)
* Patients with clinical indications for revascularization who have successfully completed percutaneous coronary intervention (PCI) prior to study enrollment

Exclusion Criteria:

* Ineligible for diagnostic IVUS examination
* Prior coronary artery bypass grafting (CABG)
* Myocardial infarction within 72 hours of coronary angiography
* Severe heart failure (NYHA grade ≥ III)
* Serum creatinine levels >150 umol/L, or glomerular filtration rates <45 ml/ kg/1.73 m2
* Allergy to the contrast agent or adenosine
* Life expectancy < 2 years
* Severe coronary artery disease requiring CABG identified during angiography
* Extreme vascular tortuosity precluding IVUS catheter advancement
* Suboptimal IVUS image quality impairing quantitative analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older admitted to Fuwai Hospital (Beijing, China) for coronary angiography and demonstrating angiographically confirmed ≥30% stenosis in all three major coronary arteries through visual assessment, will be consecutively enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 494 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) at 1 year | 1 year after the procedure
  The primary outcome is MACE at 1 year, including cardiac death, any myocardial infarction and any ischaemia-driven revascularization.

SECONDARY OUTCOMES:
Major adverse cardiac events (MACE) at 1 month | 1 month after the procedure
  MACE is defined as cardiac death, any myocardial infarction and any ischaemia-driven revascularization.
Major adverse cardiac events (MACE) at 6 months | 6 months after the procedure
  MACE is defined as cardiac death, any myocardial infarction and any ischaemia-driven revascularization.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital,Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided